CLINICAL TRIAL: NCT04652024
Title: Effect of Anorectal Biofeedback on Encopresis in School Aged Girls After Sexual Assault
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer in the deparment of pediatrics and peditaric surgery , faculty of phyical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hana4
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): Girls in the control group received pelvic floor muscle exercise (kegel exercise) daily in the outpatient clinic 12 weeks.
- STUDY GROUP (Experimental): Girls in the study group received the same physical therapy program given to the control group in addition to anorectal biofeedback for six sessions per week. in addition to kegel exercise
  Interventions: Device: Anorectal manometry

INTERVENTIONS:
Device: Anorectal manometry — , patients are instructed to isolate the anal sphincter and puborectalis muscles and improve its strength by using modified Kegel exercises in lying position with a probe in situ. Visual and verbal feedback techniques are used to reinforce the maneuvers, as they are being performed. The anal and rectal pressure changes displayed on the monitor provides visual feedback to the patient.
  Arms: STUDY GROUP

SUMMARY:
Females who have been sexually abused anally, have a disturbed anorectal motility. They have an increased resting pressure at the lower part of the anal canal. When their rectum is suddenly distended, they tend not to have an initially increased pressure in the anal canal, and the recto-anal inhibitory reflex is markedly decreased amplitude which is caused by reflex contraction of the pelvic floor during the relaxation of the internal anal sphincter.

DETAILED DESCRIPTION:
The cause of fecal incontinence after sexual abuse is the improper functioning of anal sphincter muscles, as a result of their damage and/or neurological changes including the disturbance perception of sensory stimuli from the anal canal. Biofeedback therapy using visual and verbal feedback techniques has emerged as an useful option in managing fecal incontinence and levator ani syndrome. The goal of biofeedback training is to improve bowel function by restoring a normal pattern of defecation.

ELIGIBILITY:
Inclusion Criteria:

* absent anal reflex,
* skin trifles around the anus,
* funnel shaped anus
* medically stable and able to follow instructions

Exclusion Criteria:

* sexual transmitted disease
* any medical condition that affect the anus potentially such as Crohn's disease,
* severe chronic constipation,
* myotonic dystrophy

Ages: 5 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
anorectal manometrey | pre and after 3 months of intervention, increase in the change in the mean of initial parameters of the anal and squeeze pressure indicate improvement while decreases in the mean of first sensation and maximum tolerable volume indicate improvement
  measure four variables, anal squeeze and resting pressure , first sensation and maximum tolarble volume

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa, Cairo, Egypt